CLINICAL TRIAL: NCT01978366
Title: An Open Label Extension Study of HT-100 in Patients With Duchenne Muscular Dystrophy Who Have Completed Protocol HALO-DMD-01
Brief Title: Open Label Extension Study of HT-100 in Patients With DMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dosing stopped
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO-DMD-02; HALO (Other: Akashi Therapeutics)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2019-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; halofuginone hydrobromide; anti-fibrotic; anti-inflammatory; muscle regeneration; protein synthesis inhibitor
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: HT-100 tablet, Dose 1 (Experimental): • Multiple dose administration: Dose 1
  Interventions: Drug: HT-100
- Cohort 2: HT-100 tablet, Dose 2 (Experimental): • Multiple dose administration: Dose 2
  Interventions: Drug: HT-100
- Cohort 3: HT-100 tablet, Dose 3 (Experimental): • Multiple dose administration: Dose 3
  Interventions: Drug: HT-100
- Cohort 4: HT-100 tablet, Dose 4 (Experimental): • Multiple dose administration: Dose 4
  Interventions: Drug: HT-100
- Cohort 5: HT-100 tablet, Dose 5 (Experimental): • Multiple dose administration: Dose 5
  Interventions: Drug: HT-100

INTERVENTIONS:
Drug: HT-100 — May be administered in either fed or fasted state
  Other Names: halofuginone hydrobromide delayed-release tablet

SUMMARY:
This study is designed to provide 6-months continuous dosing with the study medication, called HT-100, on participants who successfully completed the predecessor study (HALO-DMD-01). The main purpose of this study is to assess chronic safety, tolerability, pharmacodynamic activity (testing the drug's effect on DMD) and population pharmacokinetics (measuring how much drug is in the bloodstream) in participants with a broad spectrum of Duchenne muscular dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

* Completed both the single ascending dose (SAD) and multiple ascending dose (MAD) phases of predecessor study HALO-DMD-01
* Maintained the same corticosteroid therapy from the predecessor study HALO-DMD-01
* Ability to provide written informed consent
* Ambulatory or non-ambulatory

Exclusion Criteria:

* Recent, substantial change in use of cardiac medications or medications affecting muscle function
* Clinically significant major disease, not related to DMD
* Significantly compromised cardio-respiratory function
* History of severe allergic or anaphylactic reactions
* Prior treatment with another investigational product in past 6 months
* Inability to undergo magnetic resonance imaging (MRI)
* Current drug or alcohol abuse or prior treatment for abuse

Ages: 6 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of administration of 6 months of chronic, oral, multiple doses of HT-100 to boys with DMD. | Months 2, 4, 6, 7
  * Target Safety profile by review of adverse events (AEs)
  * Physical examination findings
  * Clinical laboratory test results
  * Other diagnostic testing

SECONDARY OUTCOMES:
Pharmacodynamic signals of HT-100 following chronic oral administration of multiple doses to boys with DMD. | Months 4, 6, 7
  * Pulmonary function
  * Motor function
  * Muscle composition
  * Biochemical and imaging markers
Pharmacokinetic plasma profile of HT-100 following chronic oral administration of multiple doses to boys with DMD. | Months 4, 6
  Halofuginone plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Escolar, MD, Study Director — AkashiTherapeutics
Locations (5):
- United States (5):
  - University of California, Davis Medical Center, Sacramento, California
  - Kennedy Krieger Institute, Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- See also: Sponsor company website — http://www.akashirx.com/